CLINICAL TRIAL: NCT05819749
Title: Expanding the Diabetes Homelessness Medication Support (D-Homes) Program to Spanish Speaking Hispanics
Brief Title: Diabetes Homelessness Medication Support Program in Spanish
Acronym: DH-Spanish
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hennepin Healthcare Research Institute (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-FY2023-556; R03DK133553 (NIH)
Record Dates: First submitted 2023-04-06; First posted 2023-04-19 (Actual); Results first posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-09

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Unstably Housed Persons; Hispanic or Latino; Homelessness
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: This will be an in-person, phone, or video based behavioral intervention. It will involve a diabetes wellness coach assisting participants to use behavioral activation and motivational interviewing to set goals related to diabetes self-care and co-morbidities or social conditions that get in the way of diabetes self-care. There will be encouragement to work on diabetes medication adherence and to address any un/under-treated behavioral health conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DH-Spanish Intervention (Experimental): Behavioral treatment by a diabetes wellness coach.
  Interventions: Behavioral: Diabetes Homelessness Medication Support Program in Spanish

INTERVENTIONS:
Behavioral: Diabetes Homelessness Medication Support Program in Spanish — There will be 10 sessions offered within 12 weeks to participants. Sessions will last 30-60 minutes. During sessions a diabetes wellness coach will use behavioral activation and motivational interviewing to get to know participants and set goals to improve diabetes care. The coach will encourage a focus on medication adherence behaviors to the extent that participants are willing. The coach will also help with resources and care coordination. The coach will also provide brief diabetes education as needed.
  Other Names: DH-Spanish; DHomes - Spanish

SUMMARY:
This single-arm trial of the Diabetes Homeless Medication Support intervention for Spanish-speaking people (n=12) will test the perception and feasibility of anticipated study procedures.

DETAILED DESCRIPTION:
This study has an overall goal to modify and pilot test a previously developed collaborative care intervention using motivational interviewing and behavioral activation alongside education and psychosocial support to improve medication adherence tailored to the experiences of people experiencing homelessness and diabetes (DH). The intervention was developed in English. This study is intended to test the modified intervention for DH who speak Spanish (DH-SH). The study team's central hypothesis is that medication adherence and diabetes self-care (and eventual glycemic control, health care use/cost) will improve with an intervention tailored to the unique context of DH-SH.

This protocol tests patient perceptions of the feasibility and acceptability of study procedures and refines the D-Homes treatment manual through test cases (n=12). The study team hypothesizes that the D-Homes manual and study procedures will be feasible and acceptable to DH-SH as measured by self-report and post-treatment interview.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 yrs or older
* Spanish-speaking
* Recent homelessness by federal definition (HEARTH ACT)

  1. Any housing instability in the last 12 mo. (includes supported housing or worry about paying rent)
  2. Significant housing instability in the last 24 mos. (includes any stay in shelter, outside, or places not meant for human habitation)
* Self-reported diagnosis of type 2 diabetes, later verified in medical record
* Plan to stay in local area or be reachable by phone for the next 16 weeks
* Willingness to work on medication adherence and diabetes self-care

Exclusion Criteria:

* Inability to provide informed consent (e.g. presence of a legal guardian, prisoners)
* Active psychosis or intoxication precluding ability to give informed consent
* Pregnant or lactating females
* Patients who choose to opt out of research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-02-22 (Actual); Study Completion 2024-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine D Vickery, MD, Principal Investigator — Hennepin Healthcare Research Institute
Locations (1):
- Hennepin Healthcare, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mayberry LS, Gonzalez JS, Wallston KA, Kripalani S, Osborn CY. The ARMS-D out performs the SDSCA, but both are reliable, valid, and predict glycemic control. Diabetes Res Clin Pract. 2013 Nov;102(2):96-104. doi: 10.1016/j.diabres.2013.09.010. Epub 2013 Sep 26. PMID 24209600
- [Background] Johnson JA, Coons SJ. Comparison of the EQ-5D and SF-12 in an adult US sample. Qual Life Res. 1998 Feb;7(2):155-66. doi: 10.1023/a:1008809610703. PMID 9523497
- [Background] Nguyen TD, Attkisson CC, Stegner BL. Assessment of patient satisfaction: development and refinement of a service evaluation questionnaire. Eval Program Plann. 1983;6(3-4):299-313. doi: 10.1016/0149-7189(83)90010-1. PMID 10267258

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Initial phone screener = 23 In person screening = 21 Excluded after in person screening = 9 for reason A1c below 7.5
Period: Overall Study
Arm/Group | DH-Spanish Intervention
Started | 12
Completed | 11
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | DH-Spanish Intervention
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Acceptability of Intervention
Description: Client Satisfaction Questionnaire, 8-item version, with a score range from 8-32, higher score indicating higher satisfaction.
Time Frame: at 16 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DH-Spanish Intervention
Number analyzed (Participants) | 11
score on a scale | 30.5 (0.34)

2. Secondary Outcome: Change in Glycemic Control
Description: We will measure glycemic control using hemoglobin A1c. This will be done on a consistent, validated point-of-care machine using blood samples collected via venipuncture. We will compare glycemic control from baseline to 16 weeks.
Time Frame: Baseline and 16 weeks
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Arm/Group | DH-Spanish Intervention
Number analyzed (Participants) | 11
percentage of HbA1c
  Baseline | 9.1 (1)
  16 weeks | 8.2 (1.6)

3. Secondary Outcome: Health-related Quality of Life
Description: As measured by the 12 Item Short Form Survey (SF-12), a 12-question questionnaire. The SF-12 is analyzed for two summary scores - the physical component score (PCS-12) and the mental component score (MCS-12). The average score of each component is 50 for people in the United States, with a standard deviation of 10 points. Scores above 50 indicate higher than average health-related quality of life while scores below 50 indicate lower than average health-related quality of life.
Time Frame: Baseline and 16 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DH-Spanish Intervention
Number analyzed (Participants) | 11
score on a scale
  Baseline - PCS12 | 41.2 (7.3)
  16 weeks - PCS12 | 39.7 (7.0)
  Baseline - MCS12 | 46.4 (7.7)
  16 weeks - MCS12 | 49.7 (9.1)

4. Secondary Outcome: Diabetes Medication Adherence
Description: As measured by the Adherence to Refills and Medications Scales-Diabetes (ARMS-D), Total scores range from 12-48, with higher values indicating worse outcomes. We will compare ARMS-D scores from baseline to 16 weeks.
Time Frame: Baseline and 16 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DH-Spanish Intervention
Number analyzed (Participants) | 11
score on a scale
  Baseline | 14.6 (4.3)
  16 weeks | 14.2 (4.9)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for the entire 16 weeks of each participant's involvement in the study.
Arm/Group | DH-Spanish Intervention
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-08-21): https://cdn.clinicaltrials.gov/large-docs/49/NCT05819749/Prot_SAP_000.pdf
  • Informed Consent Form (2023-04-24): https://cdn.clinicaltrials.gov/large-docs/49/NCT05819749/ICF_001.pdf